CLINICAL TRIAL: NCT03635450
Title: A Phase I Study of hCT-MSC, an Umbilical Cord-Derived Mesenchymal Stromal Cell Product, in Newborn Infants With Moderate or Severe Hypoxic- Ischemic Neonatal Encephalopathy.
Brief Title: Study of hCT-MSC in Newborn Infants With Moderate or Severe HIE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: Duke Clinical and Translational Science Institute (CTSI), part of the NIH Clinical and Translational Science Awards (CTSA) (Unknown)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor Department of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100253
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Moderate to Severe Hypoxic-ischemic Encephalopathy
Keywords: hypoxic-ischemic encephalopathy; newborn infants; therapeutic hypothermia; hCT-MSC, an Umbilical Cord Tissue-Derived Mesenchymal Stromal Cell Product
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Intervention Model Description: The first cohort of three patients will receive a single dose in the first 48 postnatal hours. If there are no safety concerns, the second cohort of three patients will receive two doses, with the first dose given in the first 48 postnatal hours and the second dose given approximately two months after the first dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First cohort of 3 subjects enrolled (Experimental): The first cohort of three patients will receive a single dose in the first 48 postnatal hours.
  Interventions: Biological: Infusion of hCT-MSC
- Second cohort of 3 subjects enrolled (Experimental): If there are no safety concerns after the first cohort of 3 subjects are infused then the second cohort of three patients will receive two doses, with the first dose given in the first 48 postnatal hours and the second dose given approximately two months after the first dose.
  Interventions: Biological: Infusion of hCT-MSC

INTERVENTIONS:
Biological: Infusion of hCT-MSC — Infants who meet enrollment criteria for moderate to severe hypoxic ischemic encephalopathy will receive 1 infusion of hCT-MSC within the first 48 postnatal hours. hCT-MSCs are a product of allogeneic cells manufactured from digested umbilical cord tissue that is expanded in culture, cryopreserved and banked. hCT-MSCs are manufactured from umbilical cord tissue donated to the Carolinas Cord Blood Bank, an FDA-licensed, FACT-accredited, public cord blood bank at Duke University Medical Center, after written informed consent from the baby's mother. Cord tissue is harvested from the placentas of male babies delivered by elective C-section after a normal, full- term pregnancy.

SUMMARY:
To determine the safety of single and repeated intravenous doses of hCT-MSC in newborn infants with HIE.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety of one and two intravenous infusions of human umbilical cord tissue-derived mesenchymal stromal cells (hCT-MSC), the first administered in the first 48 postnatal hours, and the second at two months postnatal age, in term and near term infants with moderate to severe neonatal hypoxic-ischemic encephalopathy (HIE). This is a phase I, prospective, open-label trial designed to assess the safety of one or two intravenous doses of hCT-MSC in newborn infants with moderate to severe HIE who are recipients of therapeutic hypothermia. Infants born at 36 0/7 weeks gestation or later who have moderate to severe hypoxic-ischemic encephalopathy and are receiving therapeutic hypothermia will be eligible to participate. Investigators project an accrual of 6 patients. All infants will receive intravenous infusion(s) of hCT-MSCs. The first cohort of three infants will receive a single dose in the first 48 postnatal hours. If there are no safety concerns, the second cohort of three infants will receive two doses, with the first dose given in the first 48 postnatal hours and the second dose given approximately two months after the first dose.

The potential risks associated with infusion of MSCs include a reaction to the product (rash, shortness of breath, wheezing, difficulty breathing, hypotension, swelling around the mouth, throat or eyes, tachycardia, diaphoresis), transmission of infection, and HLA sensitization. Another risk of this study is loss of confidentiality or privacy. Every effort will be made to keep the infant's medical record confidential. The results will be summarized using descriptive statistics and statistical testing as appropriate. Continuous secondary endpoints will be summarized using mean, standard deviation, CV%, median, minimum, and maximum.

ELIGIBILITY:
Inclusion Criteria:

* 36 0/7th weeks gestation or older at the time of delivery.
* Able to receive one dose of hCT-MSCs in the first 48 postnatal hours
* Willingness to return for one year assessments.
* Signs of encephalopathy within 6 hours of age

Exclusion Criteria:

* Major congenital or chromosomal abnormalities
* Severe growth restriction (birth weight <1800 g)
* Opinion by attending neonatologist that the study may interfere with clinical treatment or safety of subject
* Moribund neonates for whom no further treatment is planned
* Infants whose mothers have unknown serologies for Hepatitis B or HIV
* Infants born to mothers are known to be HIV, Hepatitis B, Hepatitis C or who have active syphilis or CMV infection in pregnancy
* Infants suspected of overwhelming sepsis
* ECMO initiated or likely in the first 48 hours of life
* Mother suspected to have intraamniotic infection at time of birth.
* ALL blood gases (cord and postnatal) done within the first 60 minutes had a pH > 7.15 AND base deficit < 10 mEq/L (source can be arterial, venous or capillary)
* Mother with documented Zika infection during this pregnancy
* Availability of autologous cord blood collected and usable in the randomized trial of autologous volume- and red blood cell-reduced cord blood cells (Duke IRB Pro00066647; clinical trials.gov link: https://clinicaltrials.gov/ct2/show/NCT02612155 )

Ages: 0 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Incidence of infusion reactions | 24 hours after each infusion
  for this study, infusion reactions are defined as anaphylactic or anaphylactoid reactions with clinical signs inclusive of skin rashes, bronchospasm, angioedema, myocardial infarcts, arrhythmias, and acute lung injury.
Incidence of Infections post-infusion | Up to 2 Weeks
  for this study, infections recorded as safety endpoints will be defined as bacterial, viral or fungal infections identified by culture or molecular methodologies within two weeks after administration of hCT-MSC.

SECONDARY OUTCOMES:
Survival | Up to 6 months
  Death prior to discharge from initial hospitalization
Neurodevelopmental Assessments | Up to 16 postnatal months
  1 year (12 - 16 postnatal months) Bayley Scales of Infant and Toddler Development, Third Edition (Bayley III) assessments in cognitive, language and motor development. Moderate to Severe CP will be assigned with cognitive score ,70, motor score ,70 and with Gross Motor Function Classification System >=2.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cotten, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No